CLINICAL TRIAL: NCT07025538
Title: Biomarker-Guided Feasibility/Efficacy Trial of Ruxolitinib in Patients With High-Risk of Chronic Graft-Versus-Host Disease Development After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Biomarker-Guided Ruxolitinib for the Prevention of Chronic Graft Versus Host Disease After Allogeneic Hematopoietic Cell Transplantation
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: budget
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24752; NCI-2025-03045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24752 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-05-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ruxolitinib) (Experimental): Starting between days +105 and +130 post-HCT, patients receive ruxolitinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo additional blood sample collection throughout the trial.
  Interventions: Other: Biomarker Analysis; Procedure: Biospecimen Collection; Other: Questionnaire Administration; Drug: Ruxolitinib
- Arm II (SOC treatment) (Active Comparator): Starting between days +105 and +130 post-HCT, patients receive SOC treatment for up to 1 year in the absence of disease progression or unacceptably toxicity. Patients also undergo additional blood sample collection throughout the trial.
  Interventions: Other: Best Practice; Other: Biomarker Analysis; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC treatment
  Other Names: standard of care; standard therapy
  Arms: Arm II (SOC treatment)
Other: Biomarker Analysis — Undergo GHVD biomarker analysis
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Ancillary studies
Drug: Ruxolitinib — Given PO
  Other Names: INCB 018424; INCB-018424; INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
  Arms: Arm I (ruxolitinib)

SUMMARY:
This phase I trial studies how well biomarker-guided ruxolitinib works for the prevention of chronic graft versus host disease (GVHD) in patients that have undergone allogeneic hematopoietic cell transplant (HCT). Allogeneic HCT is the most effective therapy for patients with high-risk blood and bone marrow malignancies. GVHD is a disease caused when cells from a donated stem cell graft attack the normal tissue of the transplant patient. Symptoms include jaundice, skin rash or blisters, a dry mouth, or dry eyes. In chronic GVHD (cGVHD), symptoms occur more than three months after transplantation. Despite significant advances in how allogeneic HCTs are conducted, cGHVD remains a major limitation to the long-term success of the transplant and can impact patients' quality of life post-transplant. Checking GVHD biomarkers in patients' blood after allogeneic HCT may help doctors predict how likely the patient is to develop cGVHD. This information can be used to help guide patients with high levels to receive cGVHD preventative therapy with ruxolitinib. Ruxolitinib works by blocking some of the enzymes that are needed for the development of cGVHD, which may be an effective way to prevent cGVHD in patients with high levels of GVHD biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of ruxolitinib administration in patients with elevated levels of chronic GVHD biomarkers at day +100 after allogeneic hematopoietic cell transplantation (HCT). (Safety lead-in) II. Evaluate the efficacy of ruxolitinib in preventing chronic GVHD by assessing 1-year moderate-to-severe cGVHD-free survival (CGFS) defined as first occurrence of moderate to severe chronic GVHD or death, whichever occurs first, after the first dose of ruxolitinib. (Expansion cohort)

SECONDARY OBJECTIVES:

I. Assess the overall survival (OS) at 1 and 2 years from enrollment and immunosuppression-free survival at 1-year from enrollment.

II. Estimate cumulative incidence of relapse and non-relapse mortality (NRM) at 1 and 2 years from enrollment.

III. Cumulative incidence and grading of chronic GVHD of all grades and moderate-to severe at 1 and 2 years from enrollment.

IV. Preliminary estimate of chronic GVHD-free and relapse-free (CRFS) at 1-year post-enrollment.

V. Cumulative incidence of severe infections requiring hospitalization at 1 and 2 years from enrollment.

VI. Quality of life assessment using Patient-Reported Outcomes Measurement Information System Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT).

VII. Further evaluation of safety of ruxolitinib for chronic GVHD prophylaxis. (Patients in the expansion cohort who are taking ruxolitinib only)

EXPLORATORY OBJECTIVES:

I. Assess levels of chronic GVHD biomarkers and other inflammatory cytokines at 6 months and 1-year post-HCT and correlate elevated levels of serum/plasma biomarkers of chronic GVHD with pre-HCT risk factors for GVHD and subsequent development of GVHD.

II. Longitudinal evaluation of the presence and levels of T cells and other immune cell subsets.

III. Assess changes in microbiome from the time of screening to 3 months after enrolment and at the time of cGVHD diagnosis.

OUTLINE: Patients undergo blood sample collection and GHVD biomarker analysis on day +100 post-HCT. Patients with elevated levels of GVHD biomarkers are assigned to arm I and patients with low levels of GVHD biomarkers are assigned to arm II.

ARM I: Starting between days +105 and +130 post-HCT, patients receive ruxolitinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo additional blood sample collection throughout the trial.

ARM II: Starting between days +105 and +130 post-HCT, patients receive standard of care (SOC) treatment for up to 1 year in the absence of disease progression or unacceptably toxicity. Patients also undergo additional blood sample collection throughout the trial.

After completion of study treatment, patients in arm I are followed up at 30 days, months 15, 18, and 24, and at the time of cGVHD diagnosis, if applicable. Patients in arm II are followed up at months 18 and 24 and at the time of cGVHD diagnosis, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* PRE-SCREENING: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* PRE-SCREENING: Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* PRE-SCREENING: Age: ≥ 18 years
* PRE-SCREENING: Karnofsky performance status ≥ 80
* PRE-SCREENING: Patients must have undergone allogeneic hematopoietic cell transplantation with peripheral blood stem cells as graft source. Note: Patients receiving manipulated graft are not included
* PRE-SCREENING: Morphologic remission per day +30 bone marrow
* PRE-SCREENING: Any conditioning regimen (myeloablative, reduce intensity/non-myeloablative conditioning) is allowed
* PRE-SCREENING: Any GVHD prophylaxis (tacrolimus-sirolimus, tacrolimus-methotrexate, or post-transplant cyclophosphamide) is allowed
* PRE-SCREENING: Life expectancy of more than 6 months
* PRE-SCREENING: Absolute neutrophil count (ANC) > 1000/mm^3 (to be performed between day +70 and +100 after HCT unless otherwise stated)
* PRE-SCREENING: Hemoglobin ≥ 8.0 gm/dL (to be performed between day +70 and +100 after HCT unless otherwise stated)
* PRE-SCREENING: Platelets ≥ 50,000/mm^3 (to be performed between day +70 and +100 after HCT unless otherwise stated)

  * Note: Patients with lower counts can enroll if infection cytomegalovirus (CMV)/human herpesvirus 6 (HHV6), etc. is being treated actively
* PRE-SCREENING: Total bilirubin ≤ 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (to be performed between day +70 and +100 after HCT unless otherwise stated)
* PRE-SCREENING: Aspartate aminotransferase (AST) =< 3.0 x ULN (to be performed between day +70 and +100 after HCT unless otherwise stated)
* PRE-SCREENING: Alanine aminotransferase (ALT) =< 3.0 x ULN (to be performed between day +70 and +100 after HCT unless otherwise stated)
* PRE-SCREENING: Glomerular filtration rate (GFR) ≥ 50 ml/min (to be performed between day +70 and +100 after HCT unless otherwise stated)
* PRE-SCREENING: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (to be performed between day +70 and +100 after HCT unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* PRE-SCREENING: Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Elevated serum/plasma levels of ST2, CXCL9, MMP-3, and OPN as indicated by moderate or severe risk of chronic GVHD in the test results
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): No use of ruxolitinib or other Jak inhibitors in the past 14 days
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Morphologic remission per day +100 bone marrow
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Adequate hematopoietic recovery (hemoglobin [Hgb] ≥ 8 g/dL, platelets [PLT] ≥ 50K/ mm^3)
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Negative serum or urine pregnancy test (female participants with childbearing potential only)
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Absence of active infection not responding to antibiotics
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Absence of progressive acute GVHD. Note: prednisone administration (flat dose of < 0.25 mg/kg) is allowed. Patients receiving any other medication to control active/progressive GVHD will be excluded
* AFTER DAY +100 TEST RESULTS PATIENTS WITH MODERATE TO HIGH-RISK cGVHD (TREATMENT ARM): Absence of any clinically significant uncontrolled sickness
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Low serum/plasma levels of ST2, CXCL9, MMP-3, and OPN as indicated by low risk of chronic GVHD in the test results
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): No use of ruxolitinib or other Jak inhibitors in the past 14 days
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Morphologic remission per day +100 bone marrow
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Adequate hematopoietic recovery (Hgb ≥ 8 g/dL, PLT ≥ 50K/ mm^3)
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Negative serum or urine pregnancy test (female participants with childbearing potential only)
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Absence of active infection not responding to antibiotics
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Absence of progressive acute GVHD. Note: prednisone administration (flat dose of < 0.25 mg/kg) is allowed. Patients receiving any other medication to control active/progressive GVHD will be excluded
* AFTER DAY +100 TEST RESULTS PATIENTS WITH LOW-RISK cGVHD (CONTROL ARM): Absence of any clinically significant uncontrolled sickness

Exclusion Criteria:

* PRE-SCREENING: Prior chemotherapy < 14 days prior to study biospecimen collection on day +100 post-HCT
* PRE-SCREENING: Previous use of ruxolitinib or other JAK-inhibitors is allowed but administration should be stopped for at least 14 days prior to enrollment. Note: Previous use of Jak inhibitors before enrollment (including the pre-HCT period) should be recorded
* PRE-SCREENING: History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* PRE-SCREENING: Active/progressive acute GVHD at the time of screening. Prednisone administration (flat dose of < 0.25 mg/kg) is allowed. Patients receiving any other medication to control active/progressive GVHD will be excluded
* PRE-SCREENING: Patients with history of major adverse cardiovascular event (MACE)/other thrombosis (myocardial infarction [MI]/stroke and pulmonary embolism [PE]/deep vein thrombosis [DVT]) in the past 6 months
* PRE-SCREENING: Patients with a history of tuberculosis
* PRE-SCREENING: Clinically significant uncontrolled illness
* PRE-SCREENING: Active infection not responding to antibiotics
* PRE-SCREENING: Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* PRE-SCREENING: Females only: Pregnant or breastfeeding
* PRE-SCREENING: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* PRE-SCREENING: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2029-06-22 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of unacceptable toxicity (UT) (Safety lead-in segment) | From first dose of ruxolitinib to end of first cycle (Cycle length = 28 days)
  UT in a given patient will be defined as any of the following that are assigned an attribution level of at least possibly related to ruxolitinib administration. 1) Any grade 3 or higher non-hematological adverse events, per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 toxicity criteria that last more than 5 days. 2) Prolonged myelosuppression, defined as ≥ grade 4 neutropenia or thrombocytopenia that persists for more than 7 days. 3) Hy's law cases. 4) Any other regimen-related cause of death. 5) Permanent discontinuation or dose reduction of ruxolitinib due to any drug-related toxicity (regardless of grade). In addition, septic UT is defined as: any grade 5 sepsis-related toxicity that is assigned an attribution level of at least possibly related to the addition of ruxolitinib to the conditioning regimen.
Chronic graft versus host disease (cGVHD) (Expansion cohort) | Up to 1 year post first dose of ruxolitinib
  Will be evaluated and scored according to National Institutes of Health (NIH) Consensus Staging.
Moderate-to-severe cGVHD free survival (GFS) | From date of starting first dose of ruxolitinib to first occurrence of moderate-to-severe cGVHD or death, whichever occurs first, assessed up to 12 months post first dose of ruxolitinib
  GFS will be censored at the last follow-up if patients are alive and remain free of moderate-to-severe cGVHD. GFS will be assessed in both the safety lead-in segment and expansion cohort. Will be analyzed using the Kaplan-Meier curves.
Patients completing at least 80% of planned ruxolitinib (Feasibility) (Expansion cohort) | Up to 1 cycle of ruxolitinib (Cycle length = 28 days)
  Patients who take at least one dose of ruxolitinib will be evaluable for feasibility. The point estimate and exact 95% confidence intervals (CIs) will be provided.
Tolerability of ruxolitinib (Expansion cohort) | Up to 12 cycles (Cycle length = 28 days)
  Patients who have ruxolitinib dose interruption, reduction, or early stopping due to adverse events attributable to ruxolitinib are deemed to be intolerable to ruxolitinib.

SECONDARY OUTCOMES:
Overall survival | From enrollment to death, assessed at 1 and 2 years post-enrollment
  Will be evaluated in all patients (those who receive ruxolitinib as pre-emptive therapy and those who did not receive ruxolitinib due to low levels of blood biomarkers). Patients are considered a failure for this endpoint if they die, regardless of cause. Will be censored at last follow-up if the last known status is alive. Will be analyzed using the Kaplan-Meier curves.
Immunosuppression-free survival | From the date of enrollment to the date of death, use of immunosuppressive agents, whichever occurs first, assessed at 1 year post-enrollment
  Patients are considered failure to this endpoint if they die (regardless of cause) or need immunosuppression (for any reason including acute or cGVHD development). Immunosuppression-free survival will be censored at last follow-up if the last known status is alive and free of immunosuppression drug usage. Will be analyzed using the Kaplan-Meier curves.
Relapse | From day of enrollment to first observation of disease relapse/progression, assessed at 1 and 2 years post-enrollment
  Deaths without relapse/progression are considered a competing risk event. Surviving patients with no history of relapse/progression are censored at time of last follow-up. Will be analyzed using the Kaplan-Meier curves.
Non-relapse mortality | From date of stem cell infusion until non-disease related death, assessed at 1 and 2 years post-enrollment
  Non-relapse mortality is defined as death occurring in a patient from causes other than relapse or progression. Will be censored at last follow-up if patients are alive and remain disease free. Will be analyzed using the Kaplan-Meier curves.
cGVHD | From day 100 through 1-year and 2- years post-transplant
  Will be evaluated and scored according to NIH Consensus Staging. The first day of cGVHD onset will be used to calculate the cumulative incidence.
cGVHD-free and relapse-free survival (CRFS) | From enrollment to cGVHD requiring systemic treatment, relapse, or death (from any cause), whichever occurs first, assessed at 1-year post-transplant
  If a patient has not experienced any of these events, CRFS is censored at the time of last follow-up. Will be analyzed using the Kaplan-Meier curves.
Incidence of infections | Up to 2 years post-enrollment
  Microbiologically documented severe infections requiring hospitalization will be reported by site of disease, date of onset, severity and resolution, if any. Tables will be constructed to summarize the observed incidence of infections. Point estimates and corresponding exact 95% CIs will be provided for each measure of infection.
Quality of life assessment _Baseline | At baseline
  Quality of life will be assessed using Patient Reported Outcomes Measurement Information System.
Quality of life assessment_3 months | 3 months post-ruxolitinib
  Quality of Life will be evaluated using the 30-item Patient-Reported Outcomes Measurement Information System (PROMIS) scale. Each item is generally rated on a 4-point Likert scale ranging from 0 (Not at all) to 4 (Extremely bothersome).Information System.
Quality of life assessment_12 months | 12 months post-ruxolitinib
  Quality of Life will be evaluated using the 30-item Patient-Reported Outcomes Measurement Information System (PROMIS) scale. Each item is generally rated on a 4-point Likert scale ranging from 0 (Not at all) to 4 (Extremely bothersome).
Quality of life assessment_24 months | 24 months post-ruxolitinib
  Quality of Life will be evaluated using the 30-item Patient-Reported Outcomes Measurement Information System (PROMIS) scale. Each item is generally rated on a 4-point Likert scale ranging from 0 (Not at all) to 4 (Extremely bothersome).
Incidence of toxicity (Ruxolitinib expansion cohort) | Up to 30 days after last dose of ruxolitinib
  Highest grades toxicities will be recorded using the NCI CTCAE v5.0 scale. Only ≥ grade 3 toxicities that are considered at least possibly related to the ruxolitinib treatment will be collected. Tables will be constructed to summarize the observed incidence, severity, and type of toxicity, including, but not limiting infections, other adverse events of special interest, and severe adverse events. Point estimates and corresponding exact 95% CIs will be provided for each measure of toxicity/adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States